CLINICAL TRIAL: NCT04609137
Title: EARLY-DIST - Early Drain Removal Versus Standard Drain Management After Distal Pancreatectomy: a Randomized Controlled Trial
Brief Title: Early Drain Removal Versus Standard Drain Management After Distal Pancreatectomy (Early-Dist)
Acronym: Early-Dist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Falconi, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Early-Dist
Record Dates: First submitted 2020-10-15; First posted 2020-10-30 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pancreas Disease; Complication,Postoperative; PROMs; Pancreatic Fistula
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Diseases; Postoperative Complications; Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early drain removal (Experimental): Participants will have an early drain removal (before postoperative day 3 (POD 3)) if specific conditions will be verified
  Interventions: Procedure: Early drain removal
- Standard drain removal (Active Comparator): Participants will receive the current standard of care at San Raffaele Hospital.
  Interventions: Procedure: Standard drain removal

INTERVENTIONS:
Procedure: Early drain removal — Patients randomized to the experimental group, will have an early drain removal if DFA on POD1 is lower than 2000 U/L and/or the drain fluid does not appear "sinister" (i.e. varying from dark brown to greenish fluid to milky water to clear "spring water" pancreatic juice like appearance) according to the clinical team. If DFA is greater than 2000 U/L, the drain will be maintained in place. If the sample on POD1 DFA is not available (e.g. drainage fluid is viscous and amylase value cannot be evaluated) or the sample could not be analyzed DFA will be evaluated on POD2, and drain removal will be considered if DFA is lower than 2000 U/L. If DFA on POD 3 is lower than 300 U/L, that is 3-fold the upper limit of normal serum amylase value, and/or the drain fluid does not appear "sinister" according to the clinical team, the drain will be removed. Otherwise, the drain will be kept in place and the patient will then follow standard postoperative drain management.
  Arms: Early drain removal
Procedure: Standard drain removal — Patients randomized to this group will receive the current standard of care, thus the drain will be maintained at least until postoperative day 5. If DFA on POD 5 is lower than 3-fold the upper limit of normal serum amylase value, and/or the drain fluid does not appear "sinister" (i.e. varying from dark brown to greenish fluid to milky water to clear "spring water" pancreatic juice like appearance) according to the clinical team, the drain will be removed. If the drain is maintained in place beyond POD 5, it will be removed inhospital or after discharge when the daily amount is lower than 10 ml and there are no signs of ongoing infection
  Arms: Standard drain removal

SUMMARY:
Main indications for distal pancreatectomy (DP) are pancreatic body and tail tumors including ductal adenocarcinoma, neuroendocrine tumors, and cystic neoplasms. Despite a less invasive operation with lower morbidity compared to pancreatic head surgery, DP is burdened by the occurrence of clinically-relevant postoperative pancreatic fistula (CR-POPF) in a significant proportion of patients.

Drain fluid amylase (DFA) on POD 1 (postoperative day 1) > 2,000 U/L appears as the best performing threshold to predict the occurrence of CR-POPF after distal pancreatectomy. Although there is preliminary evidence that early drain removal in the subgroup of patients with DFA1 < 2,000 U/L may reduce POPF, no prospective study has yet evaluated the impact of an early drain removal strategy compared to standard management.

The research question of this study is to evaluate to what extent early postoperative drain removal according to a validated DFA1 impact on clinically-relevant POPF rate after distal pancreatectomy in comparison to standard drain management. The primary hypothesis is that, early drain removal will result in a reduced proportion of patients experiencing grade B-C POPF according to ISGPS definition.

The proposed study is a two-group, assessor-blind, randomized trial. Participants will be randomly assigned with a 1:1 ratio into one of two groups: (1) standard drain management or (2) early drain removal strategy.

In this study adults (>18 years) patients with pancreatic body or tail diseases planned for distal pancreatectomy with or without splenectomy will be enrolled.The primary outcome is the POPF at 90 days after surgery, defined as grade B or C POPF according to ISGPS definition.

Participants will be asked to complete some questionnaires in order to assess their general health status, and they will be evaluated at time of hospital admission, at 15 days, at 30 days after surgery (via telephone follow-up), and at 90 days after surgery (via telephone follow-up).

DETAILED DESCRIPTION:
RATIONALE AND RESEARCH QUESTION Distal pancreatectomy (DP) is defined as the resection of the left portion of the pancreas extending from the neck to the tail of the gland. DP is burdened by the occurrence of clinically-relevant postoperative pancreatic fistula (CR-POPF) in a significant proportion of patients.Traditionally, during DP drains were placed intraoperatively in proximity of the pancreatic stump to mitigate the potential occurrence of POPF. Postoperatively, drains were usually kept in place until a POPF was ruled out by the presence of drain fluid amylase (DFA) values lower than 3-fold the upper limit of normal serum amylase, and a non "sinister" appearance of drain fluid in accordance with the International Study Group on Pancreatic Surgery (ISGPS) definition. For this reason, drains were usually maintained in place after surgery for at least 5 - 7 days. Although there is some preliminary evidence that early drain removal in the subgroup of patients with DFA1 < 2,000 U/L, no prospective study has yet evaluated the impact of an early drain removal strategy compared to standard management. Therefore, the overall aim of this study is to contribute evidence about the effect of an early drain removal policy on postoperative outcomes following distal pancreatectomy.

The primary research question is to evaluate to what extent does early postoperative drain removal according to a validated DFA1 impact on clinically-relevant POPF rate after distal pancreatectomy in comparison to standard drain management. The primary (confirmatory) hypothesis is that, early drain removal will result in a reduced proportion of patients experiencing grade B-C POPF according to ISGPS definition.

Furthermore the exploratory hypotheses that, in comparison to standard care, early drain removal will: (1) reduce time to postoperative functional recovery, (2) reduce number and severity of postoperative complications, (3) reduce postoperative surgical site infections, (4) improve self-reported physical function status, (5) improve generic health-related quality of life and (6) be cost-effective, will be tested.

STUDY DESIGN AND PARTICIPANTS The study is designed as a two-group, assessor-blind, randomized trial. Participants will be randomly assigned with a 1:1 ratio into one of two groups: (1) standard drain management or (2) early drain removal strategy. The intervention will be provided during hospital stay. Adult people with pancreatic body or tail diseases (i.e. pancreatic cancer, cystic neoplasms, pancreatic neuroendocrine tumors, etc.) planned for distal pancreatectomy with or without splenectomy at the San Raffaele Hospital IRCCS (HSR) will be considered for inclusion.

RECRUITMENT PROCESS

The step-by-step recruitment process is described below:

1. Patients scheduled for elective distal pancreatectomy who meet the inclusion/exclusion criteria will be informed about the study by a surgeon at their first office consultation
2. If the patient has interest in participating in the study, at the preoperative clinic visit or at the time of hospital admission, a trial investigator will discuss the study in detail with the patient
3. The potential participant or their legal representative will read the consent form. Once the informed consent is signed and the patient enrolled in the study, preoperative assessment will be undertaken

SURGICAL TECHNIQUE The standard surgical procedure for DP will be performed and will not be influenced by this study protocol. The choice of minimally invasive versus open technique will be at surgeon's discretion. As a general rule, patients with benign lesions or neuroendocrine tumors will be approached laparoscopically, while pancreatic cancer cases are discussed on an individual basis according to tumor location and vessel proximity. Splenectomy and standard lymphadenectomy will be routinely performed in cancer patients. A spleen preserving procedure with preservation of splenic vessels will be attempted only in non-neoplastic cases at surgeon's discretion. Pancreatic stump transection will be performed with a stapler in laparoscopic procedures, whereas in open procedures the pancreas will be cut using the scalpel followed by selective suturing of the pancreatic duct when visible.

To evaluate the association between pancreatic parenchymal structure and occurrence of POPF, in addition to standard pathology assessment, the pancreatic specimen will undergo a specific pathological evaluation. Haematoxylin and eosin (H&E) stained sections (between 1 and 4 for each case) of the pancreatic resection margin will be reviewed by two expert pancreatic pathologists, blinded to all clinical information. All the definitive slides will be assessed for their acinar, fat and fibrosis content as a proportion of the total surface area. Acinar, fat and fibrosis scores will then calculated for each patient so that their sum is equal to was 100%. The final score for each patient will be the result of two pathologists reached a consensus agreement by the two pathologists.on the scoring of each patient.

DRAIN MANAGEMENT

At the end of the operation, after reassessing exclusion criteria, participants will be randomized into one of two groups:

1. Standard postoperative drain management: Participants randomized to this group will receive the current standard of care at our institution. The drain will be maintained at least until postoperative day 5. If DFA on POD 5 is lower than 3-fold the upper limit of normal serum amylase value, and/or the drain fluid does not appear "sinister" (i.e. varying from dark brown to greenish fluid to milky water to clear "spring water" pancreatic juice like appearance) according to the clinical team, the drain will be removed. If the drain is maintained in place beyond POD 5, it will be removed inhospital or after discharge when the daily amount is lower than 10 ml and there are no signs of ongoing infection.
2. Early drain removal: Participants randomized to this group, will have an early drain removal (before POD 3) if DFA on POD1 is lower than 2000 U/L and/or the drain fluid does not appear "sinister" (i.e. varying from dark brown to greenish fluid to milky water to clear "spring water" pancreatic juice like appearance) according to the clinical team. If DFA is greater than 2000 U/L, the drain will be maintained in place. If the sample on POD1 DFA is not available (e.g. drainage fluid is viscous and amylase value cannot be evaluated) or the sample could not be analyzed (e.g. the fluid collection tube is lost or not sealed) DFA will be evaluated on POD2, and drain removal will be considered if DFA is lower than 2000 U/L. If DFA on POD 3 is lower than 300 U/L, that is 3-fold the upper limit of normal serum amylase value, and/or the drain fluid does not appear "sinister" (i.e. varying from dark brown to greenish fluid to milky water to clear "spring water" pancreatic juice like appearance) according to the clinical team, the drain will be removed. Otherwise, the drain will be kept in place and .the patient will then follow standard postoperative drain management as described above.

All patients will measure serum amylase and drain fluid amylase along with other routine postoperative laboratory tests on POD 1 - 3 - 5 as the current standard of care.

Furthermore, as drain fluid microbial contamination is considered to play a potential role for the POPF occurrence, a drain fluid culture for aerobic and /anaerobic microorganisms will be performed on POD1 (baseline) and POD5, in order to evaluate the predictive ability of early bacterial contamination in the abdominal fluid for clinically relevant POPF.

MEASUREMENTS AND OUTCOMES Demographic data, medical history, laboratory values and information relevant to the surgical procedure will be recorded. The main (confirmatory) outcome of interest will be the occurrence of CF-POPF at 90 days after surgery, defined as grade B or C POPF according to the 2016 ISGPS definition.

The proportion of patients discharged home without an abdominal drain represents the explanatory outcome measure. It will be evaluated at time of hospital discharge.

Time to functional recovery (TFR) will be measured by subtracting the date of surgery from the date when participants achieves standardized criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self-care and no evidence of untreated medical problems).

Postoperative complications occurring during the index admission or in a subsequent readmission, when related to surgery, will be recorded up to 90 days after surgery and graded by severity using the Dindo-Clavien classification. Additionally, the Comprehensive Complication Index will be calculated.

Postoperative morbidity at 90 days after surgery will include:

* Surgical site infections classified as superficial incisional, deep incisional or organ-space according to the definition by the Center for Disease Control and Prevention
* Post-pancreatectomy hemorrhage and delayed gastric empting as defined by the ISGPS Self-reported activity status will be measured using the Duke Activity Status Index (DASI) and Generic heath related quality of life will be measured using the Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile v2.1. These questionnaires will be completed before surgery, at 15, 30 and 90 days after surgery. Cost-effectiveness will be estimated by the ratio of differences in costs to differences in quality-adjusted life years (QALYs) between the two groups.

BLINDED ASSESSMENT An examiner blinded to the participants' treatment allocation will obtain all measures. The code for group allocation will not be revealed until all analyses are completed. The effectiveness of blinding will be estimated by asking the assessor to guess the participant's group allocation at the completion of the 90 days assessment. It is not possible to blind the participants to their group assignment.

STATISTICAL CONSIDERATIONS AND TIMELINES Recent studies carried at the HRS Division of Pancreatic Surgery showed that, when standard drain management is used, the proportion of patients developing CR-POPF is approximately 46%. Sample size requirement for the present study was estimated for an α level of 0.05 and 80% power to detect a 23% reduction in this proportion (risk ratio 0.23/0.46=0.5). According to this estimate, a sample of 66 participants per group is considered sufficient for our analysis. A sample size of 75 participants per group (total sample of 150) is targeted to account for possible dropouts. Regression models will be used to test the main hypothesis related to the superiority of early drain removal based on a reduction of CR-POPF at 90-days after surgery. The randomization list will be created with the "Block randomization" rule, in order to reduce bias and achieve balance in the allocation of participants to the two arms.

The Division of Pancreatic Surgery at HSR performs about 90 distal pancreatectomies annually. Based on previous trial experience, approximately 90% of these patients will be eligible and agree to participate. Therefore, 150 participants could be feasibly enrolled in 21 months. With an additional 90 days follow-up required for the primary outcome, the timeline for this study is 24 months.

SAFETY Previously completed studies have shown that early drain removal in patients with DFA1 values lower than a validated threshold in patients undergoing pancreatic head resection is not only safe but beneficial, as it reduces the incidence of CR-POPF and the risk of further complications due to the persistence of a foreign body

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) with pancreatic body or tail diseases planned for distal pancreatectomy with or without splenectomy

Exclusion Criteria:

* patient receiving an operation other than distal pancreatectomy (non-resective sx, total pancreatectomy)
* concomitant celiac trunk resection (i.e. Appleby procedure)
* concomitant multivisceral resection (i.e. colonic, gastric or liver resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of patients (n, %) developing a clinically-relevant pancreatic fistula (CR-POPF) | 90 days after surgery
  The main (confirmatory) outcome of interest will be the occurrence of clinically-relevant pancreatic fistula at 90 days after surgery, defined as grade B or C POPF according to the 2016 ISGPS definition

SECONDARY OUTCOMES:
Time to functional recovery (TFR) | 7 days after surgery
  TFR will be measured by subtracting the date of surgery from the date when participants achieves standardized criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self-care and no evidence of untreated medical problems)
Comprehensive Complication Index (CCI) | 90 days after surgery
  The Comprehensive Complication Index is a validated measure summarizing the complete spectrum of complications occurred and their severity in a single score ranging from 0 to 100. Minimum value is 0 (no complications), maximum value is 100 (mortality). Higher scores mean a worse outcome.
Number of patients (n, %) developing a postoperative Surgical Site Infection (SSI) | 90 days after surgery
  SSIs is classified as superficial incisional, deep incisional or organ-space according to the definition by the Center for Disease Control and Prevention (CDC).
  Superficial incisional SSI involves only skin and subcutaneous tissue of the incision.
  Deep incisional SSI involves deep soft tissues of the incision (for example, fascial and muscle layers).
  Organ/Space SSI involves any part of the body deeper than the fascial/muscle layers that is opened or manipulated during the operative procedure
Patient activity status - Duke Activity Status Index | Pre-surgey, 15 days, 30 days, 90 days
  Self-reported activity status will be measured using the Duke Activity Status Index (DASI), a brief questionnaire designed to assess physical function and predict exercise capacity (peak oxygen uptake). Participants are asked to respond whether they are able to perform 12 listed activities of various intensities (ambulation, household tasks, personal care and leisure activities). A specific score is given for each positive answer. The possible total score range from 0 to 58. 0 corresponds to no activity (worse outcome); 58 corresponds to performance of all activities (best outcome)
Generic health related quality of life - Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile version 2.1 | Pre-surgery, 15 days, 30 days, 90 days
  Generic heath related quality of life will be measured using the Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile v2.1 (PROPr), a questionnaire designed to measure self-reported physical, mental and social health and wellbeing. It contains 29 questions covering seven domains of health. All questions are ranked on a 5-point Likert Scale. Each domain (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) is then scored on a scale from 4 to 20. For negative domains (Depression, Anxiety, Pain Interference, Fatigue, Sleep Disturbance), lower scores represent better outcomes, higher scores represent worse outcomes. For postive domains (Ability to Participate in Social Roles and Activities and Physical Function), lower scores represent worse outcomes, higher scores represent better outcomes.
Number of patients (n, %) requiring an unplanned hospital readmission after discharge | 90 days after surgery
  Unplanned hospital readmission is defined as the need for hospitalization for treatment of a postoperative complications within 90 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Falconi, Professor, Principal Investigator — Ospedale San Raffaele IRCCS; Stefano Partelli, Investigator, Study Director — Ospedale San Raffaele IRCCS
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MK 4th, Lewis RS, Strasberg SM, Hall BL, Allendorf JD, Beane JD, Behrman SW, Callery MP, Christein JD, Drebin JA, Epelboym I, He J, Pitt HA, Winslow E, Wolfgang C, Vollmer CM Jr. Defining the post-operative morbidity index for distal pancreatectomy. HPB (Oxford). 2014 Oct;16(10):915-23. doi: 10.1111/hpb.12293. Epub 2014 Jun 16. PMID 24931404
- [Background] Miao Y, Lu Z, Yeo CJ, Vollmer CM Jr, Fernandez-Del Castillo C, Ghaneh P, Halloran CM, Kleeff J, de Rooij T, Werner J, Falconi M, Friess H, Zeh HJ, Izbicki JR, He J, Laukkarinen J, Dejong CH, Lillemoe KD, Conlon K, Takaori K, Gianotti L, Besselink MG, Del Chiaro M, Montorsi M, Tanaka M, Bockhorn M, Adham M, Olah A, Salvia R, Shrikhande SV, Hackert T, Shimosegawa T, Zureikat AH, Ceyhan GO, Peng Y, Wang G, Huang X, Dervenis C, Bassi C, Neoptolemos JP, Buchler MW; International Study Group of Pancreatic Surgery (ISGPS). Management of the pancreatic transection plane after left (distal) pancreatectomy: Expert consensus guidelines by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2020 Jul;168(1):72-84. doi: 10.1016/j.surg.2020.02.018. Epub 2020 Apr 2. PMID 32249092
- [Background] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661
- [Background] McMillan MT, Vollmer CM Jr. Predictive factors for pancreatic fistula following pancreatectomy. Langenbecks Arch Surg. 2014 Oct;399(7):811-24. doi: 10.1007/s00423-014-1220-8. Epub 2014 Jun 25. PMID 24962147
- [Background] Giglio MC, Spalding DR, Giakoustidis A, Zarzavadjian Le Bian A, Jiao LR, Habib NA, Pai M. Meta-analysis of drain amylase content on postoperative day 1 as a predictor of pancreatic fistula following pancreatic resection. Br J Surg. 2016 Mar;103(4):328-36. doi: 10.1002/bjs.10090. Epub 2016 Jan 21. PMID 26791838
- [Background] McMillan MT, Christein JD, Callery MP, Behrman SW, Drebin JA, Hollis RH, Kent TS, Miller BC, Sprys MH, Watkins AA, Strasberg SM, Vollmer CM Jr. Comparing the burden of pancreatic fistulas after pancreatoduodenectomy and distal pancreatectomy. Surgery. 2016 Apr;159(4):1013-22. doi: 10.1016/j.surg.2015.10.028. Epub 2015 Dec 6. PMID 26670325
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Maggino L, Malleo G, Bassi C, Allegrini V, Beane JD, Beckman RM, Chen B, Dickson EJ, Drebin JA, Ecker BL, Fraker DL, House MG, Jamieson NB, Javed AA, Kowalsky SJ, Lee MK, McMillan MT, Roses RE, Salvia R, Valero V 3rd, Velu LKP, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Identification of an Optimal Cut-off for Drain Fluid Amylase on Postoperative Day 1 for Predicting Clinically Relevant Fistula After Distal Pancreatectomy: A Multi-institutional Analysis and External Validation. Ann Surg. 2019 Feb;269(2):337-343. doi: 10.1097/SLA.0000000000002532. PMID 28938266
- [Background] Daniel F, Tamim H, Hosni M, Ibrahim F, Mailhac A, Jamali F. Validation of day 1 drain fluid amylase level for prediction of clinically relevant fistula after distal pancreatectomy using the NSQIP database. Surgery. 2019 Feb;165(2):315-322. doi: 10.1016/j.surg.2018.07.030. Epub 2018 Nov 7. PMID 30414706
- [Background] Seykora TF, Liu JB, Maggino L, Pitt HA, Vollmer CM Jr. Drain Management Following Distal Pancreatectomy: Characterization of Contemporary Practice and Impact of Early Removal. Ann Surg. 2020 Dec;272(6):1110-1117. doi: 10.1097/SLA.0000000000003205. PMID 30943185
- [Background] Yang F, Jin C, Hao S, Fu D. Drain Contamination after Distal Pancreatectomy: Incidence, Risk Factors, and Association with Postoperative Pancreatic Fistula. J Gastrointest Surg. 2019 Dec;23(12):2449-2458. doi: 10.1007/s11605-019-04155-7. Epub 2019 Feb 27. PMID 30815778
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Alonso J, Permanyer-Miralda G, Cascant P, Brotons C, Prieto L, Soler-Soler J. Measuring functional status of chronic coronary patients. Reliability, validity and responsiveness to clinical change of the reduced version of the Duke Activity Status Index (DASI). Eur Heart J. 1997 Mar;18(3):414-9. doi: 10.1093/oxfordjournals.eurheartj.a015260. PMID 9076377
- [Background] Carter R, Holiday DB, Grothues C, Nwasuruba C, Stocks J, Tiep B. Criterion validity of the Duke Activity Status Index for assessing functional capacity in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2002 Jul-Aug;22(4):298-308. doi: 10.1097/00008483-200207000-00014. PMID 12202852
- [Background] Thompson EG, Gower ST, Beilby DS, Wallace S, Tomlinson S, Guest GD, Cade R, Serpell JS, Myles PS. Enhanced recovery after surgery program for elective abdominal surgery at three Victorian hospitals. Anaesth Intensive Care. 2012 May;40(3):450-9. doi: 10.1177/0310057X1204000310. PMID 22577910
- [Background] Van Buren G 2nd, Bloomston M, Schmidt CR, Behrman SW, Zyromski NJ, Ball CG, Morgan KA, Hughes SJ, Karanicolas PJ, Allendorf JD, Vollmer CM Jr, Ly Q, Brown KM, Velanovich V, Winter JM, McElhany AL, Muscarella P 2nd, Schmidt CM, House MG, Dixon E, Dillhoff ME, Trevino JG, Hallet J, Coburn NSG, Nakeeb A, Behrns KE, Sasson AR, Ceppa EP, Abdel-Misih SRZ, Riall TS, Silberfein EJ, Ellison EC, Adams DB, Hsu C, Tran Cao HS, Mohammed S, Villafane-Ferriol N, Barakat O, Massarweh NN, Chai C, Mendez-Reyes JE, Fang A, Jo E, Mo Q, Fisher WE. A Prospective Randomized Multicenter Trial of Distal Pancreatectomy With and Without Routine Intraperitoneal Drainage. Ann Surg. 2017 Sep;266(3):421-431. doi: 10.1097/SLA.0000000000002375. PMID 28692468